CLINICAL TRIAL: NCT01499407
Title: A Randomized Trial to Compare Four Different Intracoronary Modalities to Reduce Thrombus Burden and Improve Microcirculatory Function in Patients With ST-elevation Myocardial Infarction: Rationale and Design of the COCTAIL II Study
Brief Title: Randomized Trial of Standard vs ClearWay-infused Abciximab and Thrombectomy for Myocardial Infarction
Acronym: COCTAIL II
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: CLI Foundation (Other)
Responsible Party: Principal Investigator, Francesco Prati, De., CLI Foundation
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: COCTAIL II
Record Dates: First submitted 2011-12-21; First posted 2011-12-26 (Estimated); Last update posted 2012-01-05 (Estimated); Status verified 2012-01

CONDITIONS: ST-elevation Myocardial Infarction
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Abciximab

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Standard abciximab bolus (Active Comparator)
  Interventions: Drug: Abciximab
- ClearWay-infused abciximab (Experimental)
  Interventions: Device: ClearWay RX catheter
- Thrombectomy plus ClearWay-infused abciximab (Experimental)
  Interventions: Device: ClearWay RX catheter
- Thrombectomy plus standard abciximab bolus (Active Comparator)
  Interventions: Drug: Abciximab

INTERVENTIONS:
Device: ClearWay RX catheter
  Arms: ClearWay-infused abciximab; Thrombectomy plus ClearWay-infused abciximab
Drug: Abciximab
  Arms: Standard abciximab bolus; Thrombectomy plus standard abciximab bolus

SUMMARY:
Subjects with ST-elevation myocardial infarction will be randomized, to one of the following: abciximab infusion with the ClearWay coronary catheter (C), standard abciximab infusion (A), thrombectomy followed by abciximab infusion with the ClearWay catheter (T+C), or thrombectomy followed by standard abciximab infusion (T+A). The primary objective is to demonstrate that abciximab infusion with the ClearWay catheter with or without manual thrombus aspiration (groups C or T+C) will result in a significant reduction of intra-stent thrombus formations when compared to intravenous or intracoronary abciximab with or without thrombectomy (groups A or T+A). The primary endpoint will be the number of cross sections with thrombus area >10% immediately after stent implantation as assessed with OCT. Additional angiographic, ECG, and clinical endpoints will be collected and adjudicated. This trial is currently being registered at ClinicalTrials.gov.

ELIGIBILITY:
Inclusion Criteria:

* ischemic symptoms must be present at rest and last for at least 10 minutes,
* within 6 hours from onset of chest pain,
* ECG changes will be persistent ST-segment elevation or new-onset left bundle branch block,
* cardiac markers can be either in the normal range or elevated (troponin I or T and/or creatine kinase-myocardial band upper limit of normal for the local laboratory assay),
* coronary angiogram must be obtained within 6 hours from onset of symptom,
* the culprit artery must be identified in a native vessel and must show a significant lesion indicative of local thrombosis with TIMI flow 0-2
* patients must have signed the informed consent form prior to performance of trial-related procedures.

Exclusion Criteria:

* baseline TIMI flow 3,
* tortuosity of coronary vessels that may prevent negotiation of target lesions with the devices that are required by the protocol,
* myocardial ischemia precipitated by a condition other than atherosclerotic coronary artery disease (e.g. arrhythmia, severe anemia, hypoxia, thyrotoxicosis, cocaine, severe valvular disease or hypotension),
* use of a fibrinolytic agent within 14 days prior to randomization,
* use of abciximab or any other glycoprotein IIb/IIIa inhibitor within 30 days prior to randomization,
* suspected active internal bleeding or history of hemorrhahagic diathesis,
* major surgery, biopsy of a parenchymal organ, eye surgery, or serious trauma within 6 weeks prior to randomization,
* gastrointestinal or genitourinary bleeding of clinical significance within 6 weeks prior to randomization,
* history of cerebrovascular accident (CVA) or transient ischemic attack within the previous 2 years or any CVA with a residual neurological deficit,
* administration of oral anticoagulants within 7 days prior to randomization unless prothrombin time ≤1.2 times control (or international normalized ratio ≤1.4),
* ongoing treatment with oral anticoagulant,
* known current platelet count less than 100.000 cells/µL,
* prior known intracranial neoplasm, arteriovenous malformation, aneurysm, or aneurysm repair,
* known allergy to abciximab or other murine proteins,
* known impaired renal function (estimated glomerular filtration rate <60 mL/min),
* coexistent condition associated with a limited life expectancy (e.g. advanced cancer),
* participation in any phase of another clinical research trial involving the evaluation of another investigational drug or device within 30 days prior to randomization, known positive pregnancy test for women of childbearing age.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2011-12; Primary Completion 2012-12 (Estimated); Study Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
Thrombus area | 1 week
  The primary endpoint of this trial will be the post-procedural number of cross sections with thrombus area >10% at optical coherence tomography.

CONTACTS AND LOCATIONS:
Locations (1):
- A. O. S. Giovanni Addolorata, Rome, RM, Italy

REFERENCES:
- [Derived] Prati F, Di Vito L, Ramazzotti V, Imola F, Pawlowski T, Materia L, Tavazzi L, Biondi-Zoccai G, Albertucci M. Randomized trial of standard versus ClearWay-infused abciximab and thrombectomy in myocardial infarction: rationale and design of the COCTAIL II study. J Cardiovasc Med (Hagerstown). 2013 May;14(5):364-71. doi: 10.2459/JCM.0b013e3283586fee. PMID 22929568